CLINICAL TRIAL: NCT05844306
Title: A Pilot Prospective Study of the RefleXion [18F]- FDG PET-CT Subsystem Imaging Performance in Patients With Various Malignancies
Brief Title: RefleXion PET/CT Imaging Performance in Patients With Various Malignancies
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: goals met
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22668; NCI-2023-01994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22668 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-16; First posted 2023-05-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Fluorodeoxyglucose F18; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device ([18F]-FDG PET-CT, X1 RMRS PET-CT) (Experimental): Patients receive [18F]-FDG injection and undergo SOC [18F]-FDG PET-CT on study. Patients with at least one PET avid lesion then undergo X1 RMRS PET-CT imaging-only session on study.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Other: Medical Device Usage and Evaluation; Device: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo [18F]-FDG PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Given via injection
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Medical Device Usage and Evaluation — Undergo X1 RMRS PET-CT
Device: Positron Emission Tomography — Undergo [18F]-FDG PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This clinical trial examines RefleXion Medical Radiotherapy System (RMRS) imaging to the standard of care (SOC) fludeoxyglucose F-18 ([18F]-FDG)- positron emission tomography (PET)-computed tomography (CT) imaging in patients with various cancers (malignancies). PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, [18F]-FDG. Because some cancers take up [18F]-FDG, cancer cells can be seen with PET. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. The RefleXion system is designed to facilitate delivery of biology-guided radiotherapy (BgRT). The RMRS uses PET emissions to guide radiotherapy delivery in real-time and has been studied for use with FDG (which is an agent used in standard PET-CT scans that targets glucose). Information gathered from this study may help researchers to improve PET-CT imaging on the RefleXion system. This information will be used in the future to improve planning and delivery of radiotherapy that will target (in real time) the signal released from the [18F]-FDG-PET-CT tracer. Comparing the imaging from the standard of care [18F]-FDG-PET-CT with the [18F]-FDG imaging from RMRS may help improve the quality of the imaging captured and determine if imaging can be done on the RMRS at the same time as planning for radiation therapy, which would reduce the number of scans needed to plan for radiation for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess imaging performance of the [18F]-FDG PET-CT subsystem on the X1 RMRS to detect lesions (primary and metastatic) in patients with various types of malignancies.

SECONDARY OBJECTIVE:

I. To determine the feasibility of generating a BgRT plan using X1 RMRS-acquired [18F]-FDG PET data derived from the imaging-only session at the studied dose level.

OUTLINE:

Patients receive [18F]-FDG injection and undergo SOC [18F]-FDG PET-CT on study. Patients with at least one PET avid lesion then undergo X1 RMRS PET-CT imaging-only session on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: >= 21 years
* Patients with malignancies (abdominal/pelvic/thoracic/head and neck/breast tumors) undergoing SOC [18F]-FDG PET-CT for diagnostic and/or radiotherapy planning purposes
* Patients should be scheduled for [18F]-FDG PET-CT prior to study entry

Exclusion Criteria:

* Known psychiatric or substance abuse disorder that would interfere with conduct of the study
* Patient weight exceeding the weight limit (450 pounds) outlined per X1 RMRS specifications sheet
* Lung parenchymal and bone tumors will be excluded as their imaging characteristics were evaluated in a previous study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Imaging performance of X1 RefleXion Medical Radiotherapy System (RMRS) positron emission tomography (PET)-computed tomography (CT) with the Imaging performance of the diagnostic fludeoxyglucose F-18 ([18F]-FDG) PET-CT | Up to 72 hours
  One key metric will be the percent of patients with lesions identified on standard of care (SOC) PET-CT that are not identified on X1 (false negatives if considering SOC the true standard).
  For the SOC [18F]-FDG PET-CT, the maximum standard uptake value (SUV) and the greatest dimension in centimeters will be recorded for each PET avid malignant lesion identified by the nuclear medicine radiologist. The patient's radiation oncologist will interpret the X1 PET scan for the same metrics.
  Graphical presentations will be provided to compare SOC positive lesions and X1 positive lesions, and SOC positive lesions and X1 negative lesions with regards to lesion size, lesion location (lymph nodes, soft tissue, visceral organ) and SUV uptake. Descriptive statistics will be utilized to quantify results. Mean, standard deviation, interquartile range (IQR), and range will be reported for each continuous variable. Frequency and percentage will be reported for categorical variables.

SECONDARY OUTCOMES:
Percent of cases where X1 RMRS PET data can be used to generate an acceptable biology-guided radiotherapy (BgRT) plan | Up to 72 hours
  The true positive lesions identified on the X1 PET images will be identified and used for BgRT planning. Simulated planning using the RefleXion treatment planning software will be performed, and the radiation dose to organs at risk calculated. Principal investigator will determine whether this plan is acceptable or not. The percent of cases in which RefleXion [18F]-FDG PET data led to an acceptable plan will be recorded (descriptive statistics). Descriptive statistics will be utilized to quantify results. Mean, standard deviation, IQR, and range will be reported for each continuous variable. Frequency and percentage will be reported for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States